CLINICAL TRIAL: NCT02864810
Title: A Phase 1, Open-label, Non-randomized, Single Center Study to Assess Safety, Pharmacokinetics, Biodistribution, Internal Radiation Dosimetry and Diagnostic Performance of [18F]GP1 Positron Emission Tomography in Subjects With Venous or Arterial Thromboembolism
Brief Title: Safety, Pharmacokinetics, Biodistribution, and Diagnostic Performance of [18F]GP1 PET in Thromboembolism
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Asan Foundation (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: GP1-1501
Record Dates: First submitted 2016-08-03; First posted 2016-08-12 (Estimated); Last update posted 2018-05-18 (Actual); Status verified 2018-05

CONDITIONS: Thromboembolism
MeSH Terms: conditions — Thromboembolism

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- [18F]GP1 PET/CT imaging (Experimental): Maximally 10 patients with deep vein thrombosis, pulmonary embolism, or arterial thromboembolism, respectively will be enrolled in the study (plus replacements for drop-outs).
  Intravenous injection and PET/CT scanning of [18F]GP1
  Interventions: Drug: [18F]GP1

INTERVENTIONS:
Drug: [18F]GP1 — [18F]GP1 PET/CT imaging for detecting thromboembolism
  Other Names: GP1

SUMMARY:
[18F]GP1 targets platelet GPIIb/IIIa receptor in thrombus. [18F]GP1 PET/CT imaging will noninvasively assess thrombus in whole body with good sensitivity with information of thrombus. Safety, pharmacokinetics, biodistribution, internal radiation dosimetry and diagnostic performance of [18F]GP1 will be assessed in all subjects.

ELIGIBILITY:
Inclusion Criteria:

* Patient is ≥ 19 years of age and male or female of any race/ethnicity.
* Patient has signs or symptoms of acute DVT of the leg, acute PE or ATE; or had arterial intervention or surgery, such as endovascular abdominal aortic aneurysm repair preferably within 14 days prior to the planned study with [18F]GP1.
* Patient has thromboembolic focus/foci confirmed by standard imaging modalities within 5 days prior to administration of [18F]GP1.
* Patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0-2 at time of screening.
* Patient has clinical laboratory tests that are within the following ranges, determined within 7 days prior to administration of [18F]GP1:

  * White blood cell count ≥ 3.0 x 109/L;
  * Platelets ≥ 75.0 x 109/L;
  * ALT and AST ≤ 3.0 times upper limit of normal;
  * Bilirubin ≤ 1.5 times upper limit of normal; and
  * Serum creatinine ≤ 1.5 times upper limit of normal

Exclusion Criteria:

A patient will be excluded from this study if the patient does not fulfill the inclusion criteria, or if any of the following conditions are observed:

* Patient or patient's legally acceptable representative does not provide written informed consent.
* In case of acute DVT or PE, patient has a previous history of objectively diagnosed DVT or PE.
* Patient had pretreatment with glycoprotein IIb/IIIa inhibitors within 15 days before the administration of [18F]GP1
* Chemotherapy is scheduled to given to patient before or within 24 hours after administration of [18F]GP1.
* Female patient is pregnant or nursing.
* Patient has concurrent severe and/or uncontrolled and/or unstable medical disease other than cancer (e.g. congestive heart failure, acute myocardial infarction, severe pulmonary disease, chronic renal or hepatic disease which could compromise participation in the study) in the judgment of the investigator.
* Patient is a relative of the investigator, student of the investigator or otherwise dependent.
* Patient has been involved in another investigative clinical study involving administration of an investigational drug from preceding 4 weeks before to 24 hours after administration of [18F]GP1.
* Patient has been previously included in this study.
* Patient has any other condition or personal circumstances that, in the judgment of the investigator, might make collection of complete data difficult or impossible.
* Additive-related precautions: This investigational product contains sodium bisulfite, a sulfite that may cause allergic-type reactions including anaphylactic symptoms and life-threatening or less severe asthmatic episodes in certain susceptible people. The overall prevalence of sulfite sensitivity in the general population is unknown and probably low. Sulfite sensitivity is seen more frequently in asthmatic than in nonasthmatic people.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-08-04 (Actual); Primary Completion 2017-09-09 (Actual); Study Completion 2017-09-09 (Actual)

PRIMARY OUTCOMES:
Detection rate of thromboembolic focus/foci with [18F]GP1 PET/CT | 6 months

SECONDARY OUTCOMES:
Quantitative assessment of [18F]GP1 uptake in thromboembolic focus/foci as measured by standardized uptake value (SUV) | 6 months
Biodistribution and radiation dosimetry of [18F]GP1 as measured by SUV | 6 months
Biodistribution and radiation dosimetry of [18F]GP1 as measured by radiation doses per organ (μGy/MBq). | 6 months
Pharmacokinetics of [18F]GP1 as measured by area under the curve | 6 months
Pharmacokinetics of [18F]GP1 as measured by Cmax | 6 months
Pharmacokinetics of [18F]GP1 as measured by Tmax | 6 months
Pharmacokinetics of [18F]GP1 as measured by percent fraction | 6 months
Safety of [18F]GP1 as measured by the number of participants with adverse events and significant changes in vital signs, electrocardiogram, physical examination and laboratory data that are related to treatment. | 6 months
  Evaluation of safety of [18F]GP1
Correlation of [18F]GP1 activity with fibrinogen and platelet glycoprotein IIb/IIIa and P-selectin expression. | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Foundation, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chae SY, Kwon TW, Jin S, Kwon SU, Sung C, Oh SJ, Lee SJ, Oh JS, Han Y, Cho YP, Lee N, Kim JY, Koglin N, Berndt M, Stephens AW, Moon DH. A phase 1, first-in-human study of 18F-GP1 positron emission tomography for imaging acute arterial thrombosis. EJNMMI Res. 2019 Jan 7;9(1):3. doi: 10.1186/s13550-018-0471-8. PMID 30617563